CLINICAL TRIAL: NCT00485069
Title: Post-Marketing Clinical Study of REQUIP (Ropinirole Hydrochloride) Tablets in Patients With Parkinson's Disease- Evaluation of Long-Term Efficacy and Safety -
Brief Title: REQUIP (Ropinirole Hydrochloride) IR Long-Term Phase 4 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108862
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson Disease; Parkinson's Disease
Keywords: Ropinirole hydrochloride; L-dopa; Parkinson's Disease; Dopamine agonist
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- Ropinirole Hydrochloride (Experimental)
  Interventions: Drug: ROP; Drug: ROP+L-Dopa

INTERVENTIONS:
Drug: ROP — Ropinirole Hydrochloride monotherapy group (ROP): Patients will receive ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose will start at 0.75 mg/day and will be increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose will be increased by 1.5 mg/day at intervals of at least 1 week up to a maximum of 15.0 mg/day. The dose will be maintained at a level without further symptomatic improvement is expected. Concomitant use of L-dopa is prohibited during the study.
Drug: ROP+L-Dopa — Ropinirole Hydrochloride with L-Dopa adjunct therapy group (ROP+L-Dopa): Patients will receive ropinirole hydrochloride (ROP) tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose will start at 0.75 milligrams (mg)/day and will be increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose will be increased by 1.5 mg/day at intervals of at least 1 week up to a maximum of 15.0 mg/day. The dose will be maintained at a level without further symptomatic improvement is expected. The dosing regimen of L-dopa remain unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.

SUMMARY:
Ropinirole Hydrochloride (ROP) was granted approval for the treatment of Parkinson's Disease (PD) on 20 October 2006.

ROP is expected to be used for a long term in clinical practice. However, no long-term clinical data with ROP administered three times daily are currently available from Japanese patients, and the clinical experience with ROP at >10mg/day is limited.

For this reason, this study was designed as a multicenter open-label uncontrolled study.

This study will evaluate the long-term efficacy (Japanese Unified Parkinson's Disease Rating Scale (UPDRS), Awake time spent "Off"/"On", Modified Hoehn & Yahr stage, Schwab-England scale, Proportion of subjects remaining in this study and Clinical Global Impression (CGI)) and the long-term safety of ROP administered three times daily for in PD patients.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria. Note that both inpatients and outpatients are eligible.

* Patients with a diagnosis of PD (including juvenile parkinsonism) with Modified Hoehn & Yahr Stages I to IV.
* Patients who have been receiving another dopamine agonist for at least 4 weeks prior to the start of the screening phase and are expected to benefit from conversion to ROP.
* Age: 20 years (at the time of written informed consent).
* Informed consent: Patients who are able to give written informed consent in person (i.e., patients who are capable of giving written informed consent on their own).
* Gender: Male or female

Females of childbearing potential are eligible for enrollment in the study, only if the subject has a negative pregnancy test at the start of the screening phase and agrees to conduct pregnancy testing at the protocol-specified visits during the study and use one of the following acceptable methods of contraceptions properly and accurately:

* Abstinence
* Oral contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring (Caution: This should be used cautiously, because the blood concentration of the study drug may be increased.)
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS)
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject)
* Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (foam/gel/film/cream/suppository)

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Patients who present with any serious medical condition other than PD (e.g., cardiac, hepatic or renal disorder or hematopoietic disorder).

Serious is defined as Grade 3 as a rule according to the Classification of the Severity of Adverse Experiences.

* Patients with postural hypotension with any subjective symptoms (e.g., dizziness and syncope).
* Patients who have had any serious psychiatric symptoms (e.g., confusion, hallucination, delusion, abnormal behavior) (including symptoms caused by anti-PD drugs) within 6 months (26 weeks) prior to written informed consent.
* Patients who have initiated any of the following drugs within 4 weeks of the start of the screening phase and have the dosing regimen of the drug changed within 4 weeks of the start of the screening phase.

  * L-dopa (+DCI) (NOTE: This does not apply to the monotherapy group.)
  * Anticholinergic agents: trihexyphenidyl hydrochloride, piroheptine hydrochloride, mazaticol hydrochloride, metixene hydrochloride, biperiden, profenamine
  * amantadine hydrochloride
  * droxidopa
  * citicoline
  * selegiline hydrochloride
  * entacapone
  * zonisamide
* Patients with severe dementia with a Japanese UPDRS Part I (mentation, behavior, and mood) score of 3 or 4.
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study period or within 30 days after the last dose of the study drug.
* Patients with a history of drug allergy to any ingredients of ROP tablets.
* Patients who have received surgical treatment for PD in the past (e.g., pallidectomy, deep brain stimulation).
* Patients who have been treated with any other investigational product within 12 weeks prior to the start of the screening phase.
* Patients who, in the judgement of the investigator (or sub-investigator), have evidence of alcohol or drug abuse.
* Others whom the investigator (or sub-investigator) considers ineligible for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Japan (12):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 weeks of Treatment Phase, consisting of 4 weeks of Fixed Titration Phase and 48 weeks of Flexible Titration and Maintenance Phase, was started after 1 to 4 weeks of Screening Phase. Although the results are presented by participants with and without L-dopa, this study was a single-arm design, and L-dopa was not the investigational product.
Groups:
- ROP+L-Dopa: Participants received ropinirole hydrochloride (ROP) tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 milligrams (mg)/day and was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals of at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
- Ropinirole Hydrochloride: Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day and was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals of at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. Concomitant use of L-dopa was prohibited during the study.
Period: Overall Study
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Started | 65 | 58
Completed | 47 | 46
Not Completed | 18 | 12
Not completed — Adverse Event | 10 | 4
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- ROP+L-Dopa: Participants received ropinirole hydrochloride (ROP) tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 milligrams (mg)/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
- Ropinirole Hydrochloride: Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. Concomitant use of L-dopa was prohibited during the study.
- Total: Total of all reporting groups
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride | Total
Number analyzed (Participants) | 65 | 58 | 123
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (7.94) | 65.5 (7.18) | 65.8 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 38 | 27 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 65 | 58 | 123
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Japanese Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score (in "On" State for the ROP+L-Dopa Group) at Week 52 and Final Assessment Point (FAP)
Description: The Japanese UPDRS assesses the status of Parkinson's Disease (PD) patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. Participants with "off" state at baseline or without post-baseline data were not included in the ROP+L-dopa group at FAP. These participants as well as one with "off" state at Week 52 and those prematurely withdrawn were not included at Week 52.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: Full Analysis Set (FAS): all participants enrolled in the Treatment Phase, excluding those with objective measurements not meeting the major eligibility criteria, who did not receive ROP at all, and those with no valid post-baseline data. Last observation carried forward (LOCF) was used for the FAP data to impute post-baseline missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Week 52, n=45, 46 | -7.0 (8.17) | -6.9 (7.56)
  FAP, n=61, 58 | -5.8 (8.33) | -5.5 (8.08)

2. Secondary Outcome: Mean Change From Baseline in the Japanese UPDRS Part I Total Score at Week 52 and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. One participant was not included in the ROP+L-dopa group at FAP as having no post-baseline data. This participant as well as those prematurely withdrawn from the study in each group was not included at Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ROP+L-Dopa: Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Week 52, n=47, 46 | -0.4 (1.11) | -0.1 (0.90)
  FAP, n=64, 58 | -0.2 (1.26) | -0.0 (0.96)

3. Secondary Outcome: Mean Change From Baseline in the Japanese UPDRS Part II Total Score at Week 52 and FAP by "On"/"Off" State in the ROP+L-Dopa Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. "Off" state is where PD symptoms are not adequately controlled by the drug.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Some participants were not included at FAP as having no post-baseline data in "on" state, not having "off" state at baseline, or no data in "off" state at Week 52/withdrawal. These participants as well as those prematurely withdrawn were not included at Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ROP+L-Dopa, "On" State; ROP+L-Dopa, "Off" State (Only Participants With "Off" State): Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
Arm/Group | ROP+L-Dopa, "On" State | ROP+L-Dopa, "Off" State (Only Participants With "Off" State)
Number analyzed (Participants) | 65 | 32
units on a scale
  Week 52, n=47, 13 | -3.5 (4.19) | -2.8 (3.77)
  FAP, n=64, 22 | -2.3 (4.54) | -0.3 (6.46)

4. Secondary Outcome: Mean Change From Baseline in the Japanese UPDRS Part II Total Score at Week 52 and FAP in the ROP Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Participants prematurely withdrawn from the study were not included at Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
units on a scale
  Week 52, n=46 | -2.2 (3.60)
  FAP, n=58 | -1.8 (3.86)

5. Secondary Outcome: Mean Change From Baseline in the Japanese UPDRS Part IV Total Score at Week 52 and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Week 52, n=47, 46 | 0.1 (1.54) | 0.3 (1.24)
  FAP, n=64, 58 | 0.3 (1.75) | 0.3 (1.15)

6. Secondary Outcome: Japanese UPDRS Part I Mean Total Score at Baseline, Week 52, and FAP
Description: as for outcome 2
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Baseline, n=65, 58 | 0.8 (1.35) | 0.8 (1.10)
  Week 52, n=47, 46 | 0.4 (0.77) | 0.7 (1.11)
  FAP, n=64, 58 | 0.7 (1.30) | 0.8 (1.15)

7. Secondary Outcome: Mean Percent Change From Baseline in the Japanese UPDRS Part I Total Score at Week 52 and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms. Percent change from baseline was calculated as (change from baseline score/baseline score) * 100; change from baseline was calculated as thescore at the observation day minus the baseline score.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Some participants were not included at FAP as having a baseline value of zero, which could not be used for calculating the percent change, or having no post-baseline data. These participants as well as those prematurely withdrawn in each group were not included at Week 52.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
percent change in score
  Week 52, n=19, 22 | -68.86 (41.929) | -22.73 (79.772)
  FAP, n=27, 26 | -38.09 (109.715) | -21.92 (73.595)

8. Secondary Outcome: Japanese UPDRS Part II Mean Total Score at Baseline, Week 52, and FAP by "On"/"Off" State in the ROP+L-Dopa Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. "Off" state is where PD symptoms are not adequately controlled by the drug. LOCF was used for the FAP data. Some participants were not included at FAP as having no post-baseline data in "on" state or having no data in "off" state at Week 52/withdrawal.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. Participants without "off" state at baseline were not included in the analysis of baseline "off" state data. Participants not included at FAP as well as those prematurely withdrawn from the study were not included at Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ROP+L-Dopa, "Off" Sate (Only Participants With "Off" State): Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
Arm/Group | ROP+L-Dopa, "On" State | ROP+L-Dopa, "Off" Sate (Only Participants With "Off" State)
Number analyzed (Participants) | 65 | 32
units on a scale
  Baseline, n=65, 27 | 7.9 (5.51) | 14.3 (9.04)
  Week 52, n=47, 16 | 4.1 (4.37) | 11.4 (5.93)
  FAP, n=64, 26 | 5.5 (6.18) | 15.2 (10.98)

9. Secondary Outcome: Japanese UPDRS Part II Mean Total Score at Baseline, Week 52, and FAP in ROP Group
Description: as for outcome 4
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
units on a scale
  Baseline, n=58 | 7.7 (4.59)
  Week 52, n=46 | 5.4 (4.65)
  FAP, n=58 | 5.9 (4.52)

10. Secondary Outcome: Mean Percent Change From Baseline in the Japanese UPDRS Part II Total Score at Week 52 and FAP by "On"/"Off" State in the ROP+L-Dopa Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. "Off" state is where PD symptoms are not adequately controlled by the drug. Percent change from baseline was calculated as (change from baseline score/baseline score) * 100; change from baseline was calculated as thescore at the observation day minus the baseline score.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for FAP data. Some participants were not included at FAP as having a baseline value of zero, having no post-baseline data in "on" state, not having "off" state at baseline in "off" state, or having no data at Week 52/withdrawal in "off" state. These participants as well as those prematurely withdrawn were not included at Week 52.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | ROP+L-Dopa, "On" State | ROP+L-Dopa, "Off" State (Only Participants With "Off" State)
Number analyzed (Participants) | 65 | 32
percent change in score
  Week 52, n=47, 13 | -48.98 (45.862) | -17.68 (31.381)
  FAP, n=62, 22 | -29.00 (73.391) | -4.10 (36.155)

11. Secondary Outcome: Mean Percent Change From Baseline in the Japanese UPDRS Part II Total Score at Week 52 and FAP in the ROP Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. Percent change from baseline was calculated as (change from baseline score/baseline score) * 100; change from baseline was calculated as thescore at the observation day minus the baseline score.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Some participants were not included at FAP as having a baseline value of zero, which could not be used for calculating the percent change. These participants as well as those prematurely withdrawn were not included at Week 52
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
percent change in score
  Week 52, n=44 | -24.35 (59.429)
  FAP, n=56 | -16.74 (61.175)

12. Secondary Outcome: Japanese UPDRS Part III Mean Total Score (in "On" State for the ROP+L-Dopa Group) at Baseline, Week 52, and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. LOCF was used for the FAP data to impute post-baseline missing values. One participant was not included in the ROP+L-dopa group at FAP as having no post-baseline data.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. Participants having "off" state at baseline were not included in the ROP+L-dopa group at baseline. The participant not included in the FAP as well as one having "off" state in the ROP+L-dopa group at Week 52 and those prematurely withdrawn in each group were not included at Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Baseline, n=62,58 | 20.5 (12.44) | 19.8 (12.10)
  Week 52, n=46, 46 | 12.7 (10.26) | 13.1 (10.86)
  FAP, n=64, 58 | 14.3 (12.20) | 14.3 (11.01)

13. Secondary Outcome: Mean Percent Change From Baseline in the Japanese UPDRS Part III Total Score (in "On" State for the ROP+L-Dopa Group) at Week 52 and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. "On" state is where PD symptoms are well controlled by the drug. Percent change from baseline was calculated as (change from baseline score/baseline score) * 100; change from baseline was calculated as thescore at the observation day minus the baseline score.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Participants with "off" state at baseline or without post-baseline data were not included in the ROP+L-dopa group at FAP. These participants as well as one with "off" state at Week 52 in that group and those prematurely withdrawn in each group were not included at Week 52.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
percent change in score
  Week 52, n=45, 46 | -36.83 (40.001) | -37.73 (34.739)
  FAP, n=61, 58 | -30.42 (41.427) | -27.79 (42.531)

14. Secondary Outcome: Japanese UPDRS Part IV Mean Total Score at Baseline, Week 52, and FAP
Description: as for outcome 5
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
units on a scale
  Baseline, n=65, 58 | 2.1 (3.01) | 0.5 (1.17)
  Week 52, n=47, 46 | 1.5 (1.77) | 0.8 (1.33)
  FAP, n=64, 58 | 2.4 (3.30) | 0.8 (1.26)

15. Secondary Outcome: Mean Percent Change From Baseline in the Japanese UPDRS Part IV Total Score at Week 52 and FAP
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications. Percent change from baseline was calculated as (change from baseline score/baseline score) * 100; change from baseline was calculated as thescore at the observation day minus the baseline score.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Some participants were not included at FAP as having a baseline value of zero, which could not be used for calculating the percent change, or having no post-baseline data. These participants as well as those prematurely withdrawn from the study were not included at Week 52.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
percent change in score
  Week 52, n=23, 17 | -8.70 (62.889) | 0.00 (115.920)
  FAP, n=37, 20 | 13.30 (91.068) | -2.50 (109.394)

16. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Scale at Baseline, Week 52, and FAP by "On"/"Off" State in the ROP+L-Dopa Group
Description: The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided. LOCF was used for the FAP data to impute post-baseline missing values. Some participants in each state were not included at FAP as having no post-baseline data in the corresponding state or having no data in the corresponding state at Week 52/withdrawal.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | ROP+L-Dopa, "On" State | ROP+L-Dopa, "Off" State (Only Participants With "Off" State)
Number analyzed (Participants) | 65 | 32
participants
  Baseline, n=65, 27, Stage 0 | 0 | 0
  Baseline, n=65, 27, Stage 1 | 5 | 0
  Baseline, n=65, 27, Stage 1.5 | 3 | 1
  Baseline, n=65, 27, Stage 2 | 22 | 2
  Baseline, n=65, 27, Stage 2.5 | 16 | 9
  Baseline, n=65, 27, Stage 3 | 16 | 7
  Baseline, n=65, 27, Stage 4 | 3 | 6
  Baseline, n=65, 27, Stage 5 | 0 | 2
  Week 52, n=47, 16, Stage 0 | 1 | 0
  Week 52, n=47, 16, Stage 1 | 10 | 1
  Week 52, n=47, 16, Stage 1.5 | 6 | 1
  Week 52, n=47, 16, Stage 2 | 15 | 1
  Week 52, n=47, 16, Stage 2.5 | 6 | 4
  Week 52, n=47, 16, Stage 3 | 8 | 4
  Week 52, n=47, 16, Stage 4 | 1 | 4
  Week 52, n=47, 16, Stage 5 | 0 | 1
  FAP, n=63, 25, Stage 0 | 1 | 0
  FAP, n=63, 25, Stage 1 | 13 | 1
  FAP, n=63, 25, Stage 1.5 | 7 | 1
  FAP, n=63, 25, Stage 2 | 21 | 1
  FAP, n=63, 25, Stage 2.5 | 7 | 5
  FAP, n=63, 25, Stage 3 | 11 | 7
  FAP, n=63, 25, Stage 4 | 3 | 7
  FAP, n=63, 25, Stage 5 | 0 | 3

17. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Scale at Baseline, Week 52, and FAP in the ROP Group
Description: The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided.
Time Frame: Number of Participants at Each Stage of the Modified Hoehn & Yahr Scale at Baseline, Week 52, and FAP in the ROP Group
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
participants
  Baseline, n=58, Stage 0 | 0
  Baseline, n=58, Stage 1 | 9
  Baseline, n=58, Stage 1.5 | 2
  Baseline, n=58, Stage 2 | 21
  Baseline, n=58, Stage 2.5 | 14
  Baseline, n=58, Stage 3 | 12
  Baseline, n=58, Stage 4 | 0
  Baseline, n=58, Stage 5 | 0
  Week 52, n=46, Stage 0 | 1
  Week 52, n=46, Stage 1 | 12
  Week 52, n=46, Stage 1.5 | 1
  Week 52, n=46, Stage 2 | 14
  Week 52, n=46, Stage 2.5 | 13
  Week 52, n=46, Stage 3 | 5
  Week 52, n=46, Stage 4 | 0
  Week 52, n=46, Stage 5 | 0
  FAP, n=58, Stage 0 | 1
  FAP, n=58, Stage 1 | 13
  FAP, n=58, Stage 1.5 | 2
  FAP, n=58, Stage 2 | 17
  FAP, n=58, Stage 2.5 | 18
  FAP, n=58, Stage 3 | 7
  FAP, n=58, Stage 4 | 0
  FAP, n=58, Stage 5 | 0

18. Secondary Outcome: Mean Change From Baseline in the Schwab and England Activities of Daily Living Scale Score by Clinician at Week 52 and FAP by "On"/"Off" State in the ROP+L-Dopa Group
Description: The Schwab and England Activities of Daily Living Scale Score is measured as percentage, from 100% (Completely independent. Able to do all chores without slowness, difficulty or impairment. Essentially normal. Unaware of any difficulty) to 0% (Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden).
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data. Some participants were not included at FAP as having no post-baseline data in "on" state, not having "off" state at baseline in "off" state, or having no data in the corresponding state at Week 52/withdrawal. These participants as well as those prematurely withdrawn were not included at Week 52.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ROP+L-Dopa, "On" State | ROP+L-Dopa, "Off" State (Only Participants With "Off" State)
Number analyzed (Participants) | 65 | 32
percent change
  Week 52, n=47, 13 | 3.4 (10.52) | 5.8 (16.31)
  FAP, n=63, 21 | 3.0 (9.97) | 2.6 (14.63)

19. Secondary Outcome: Mean Change From Baseline in the Schwab and England Activities of Daily Living Scale Score by Clinician at Week 52 and FAP in ROP Group
Description: as for outcome 18
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
percent change
  Week 52, n=46 | 2.1 (6.74)
  FAP, n=58 | 1.5 (7.28)

20. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days in the ROP+L-Dopa Group
Description: The percentage of participants remaining in the study was presented by Kaplan-Meier method, where premature discontinuation (i.e., withdrawal before Week 52) was the event, and participants who had completed the study were censored.
Time Frame: Days 0-422
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | ROP+L-Dopa
Number analyzed (Participants) | 65
percentage of participants
  Day 0 | 100
  Day 22 | 98
  Day 33 | 95
  Day 43 | 94
  Day 85 | 92
  Day 101 | 91
  Day 112 | 89
  Day 128 | 88
  Day 154 | 86
  Day 169 | 83
  Day 196 | 82
  Day 203 | 80
  Day 238 | 78
  Day 282 | 77
  Day 301 | 75
  Day 341 | 74
  Day 365 | 72
  Day 422 | 72

21. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days in the ROP Group
Description: as for outcome 20
Time Frame: Days 0-419
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole Hydrochloride
Number analyzed (Participants) | 58
percentage of participants
  Day 0 | 100
  Day 14 | 98
  Day 29 | 97
  Day 36 | 95
  Day 66 | 93
  Day 71 | 91
  Day 85 | 90
  Day 167 | 88
  Day 169 | 86
  Day 175 | 84
  Day 210 | 83
  Day 241 | 81
  Day 253 | 79
  Day 419 | 79

22. Secondary Outcome: Number of Participants Scored as Responders on the Clinician's Global Impression (CGI) Scale at Week 52 and FAP
Description: CGI is measured on the following 7-point scale: 1, Very much improved; 2, Much Improved; 3, Minimally improved; 4, No change; 5, Minimally worse; 6, Much worse; and 7, Very much worse. Responders are defined as those participants scored as "very much improved" or "much improved."
Time Frame: Week 52 and FAP (up to Week 52)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Number analyzed (Participants) | 65 | 58
participants
  Week 52, n=47, 46 | 33 | 28
  FAP, n=64, 58 | 34 | 31

23. Secondary Outcome: Mean Change From Baseline in Awake Time "Off" (Hours) and Awake Time "On" (Hours) at Week 52 and FAP in the ROP+L-Dopa Group Excluding Participants With "0" Off (Hour) at Baseline
Description: "Off" state is where PD symptoms are not adequately controlled by the drug. "On" state is where PD symptoms are well controlled by the drug. The "off's" duration (awake time spent "off") and the "on's" duration (awake time spent "on") on each day were calculated.
Time Frame: Baseline, Week 52, and FAP (up to Week 52)
Population: FAS. LOCF was used for the FAP data to impute post-baseline missing values. Participants having "off" hour of zero at baseline were not included at FAP. These participants as well as those prematurely withdrawn from the study were not included at Week 52.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- ROP+L-Dopa, "Off" Hours; ROP+L-Dopa, "On" Hours: Participants received ROP tablets 3 times daily. In the 4-week Fixed Titration Phase (from Week 0 as Baseline), the dose started at 0.75 mg/day was increased weekly by 0.75 mg/day up to 3.0 mg/day. In the 48-week Flexible Titration and Maintenance Phase, the dose was increased by 1.5 mg/day at intervals at least 1 week up to a maximum of 15.0 mg/day. The dose was maintained at a level without further symptomatic improvement expected. The dosing regimen of L-dopa remained unchanged from 4 weeks prior to the start of the Screening Phase throughout the study.
Arm/Group | ROP+L-Dopa, "Off" Hours | ROP+L-Dopa, "On" Hours
Number analyzed (Participants) | 65 | 65
hours
  Week 52, n=16 | -0.09 (3.502) | 1.00 (4.090)
  FAP, n=22 | -0.40 (3.453) | 1.00 (3.867)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) through the end of follow-up (up to Week 56).
Arm/Group | ROP+L-Dopa | Ropinirole Hydrochloride
Serious Adverse Events (participants affected / at risk) | 7/65 | 3/58
Other Adverse Events (participants affected / at risk) | 42/65 | 43/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ROP+L-Dopa (N=65) | Ropinirole Hydrochloride (N=58)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Parkinson's Disease (Nervous system disorders) | 1 | 0
Sudden onset of sleep (Nervous system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ROP+L-Dopa (N=65) | Ropinirole Hydrochloride (N=58)
Somnolence (Nervous system disorders) | 16 | 14
Headache (Nervous system disorders) | 4 | 3
Parkinson's Disease (Nervous system disorders) | 7 | 0
Sudden onset of sleep (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 0 | 4
Dyskinesia (Nervous system disorders) | 4 | 0
Tremor (Nervous system disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 13 | 19
Nausea (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 7 | 2
Dental caries (Gastrointestinal disorders) | 2 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Hallucination (Psychiatric disorders) | 4 | 5
Orthostatic hypotension (Vascular disorders) | 3 | 5
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.